CLINICAL TRIAL: NCT00856245
Title: Role of Rituximab Containing Salvage Chemotherapy and in Vivo Purging in Obtaining PCR Negative Leukapheresis Product in Patients With Relapsed Follicular Lymphoma or Transplant Eligible Mantle Cell Lymphoma
Brief Title: Evaluate Rituximab in Obtaining PCR (Polymerase Chain Reaction) Negative Leukapheresis Product in Patients With Relapsed Follicular Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11571
Record Dates: First submitted 2009-03-03; First posted 2009-03-05 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Non-Hodgkins Lymphoma
Keywords: non-Hodgkins; lymphoma; stem cell transplant
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rituximab (Other): Patients will be treated IV with rituximab at the rate of 50 milligrams per hour (mg/hour) for 1 hour. If patient tolerates the infusion, the rate is increased by increments of 50 mg/hour every 30 minutes to a maximum of 400 mg/hour. If patient has a severe reaction, the infusion is stopped temporarily and the infusion rate is decreased by 50%. Subsequent infusions are started at the rate of 100 mg/hour, increased by 100 mg/hour every 30 minutes to a maximum of 400 mg/hour if tolerated. Vital signs are monitored every 15 minutes for 2 hours and every 30 minutes thereafter.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — 375 MG/M2 (milligram per meter squared) given IV (intravenously) weekly x 4-8 doses.
  Other Names: Rituxan

SUMMARY:
Researchers hope to learn if adding rituximab with high doses of chemotherapy and stem cell transplantation will help patients get rid of their lymphoma cells from the bone marrow and stem cell collections.

DETAILED DESCRIPTION:
Following the first relapse, patients with follicular type of Non-Hodgkin's lymphoma may have an option to receive high dose chemotherapy followed by autologous (from you) blood stem cell transplantation. One of the common causes of relapse is persistence of lymphoma cells in the bone marrow and in the collected stem cell products.

Patients who do not have a complete response after traditional chemotherapy, have a greater chance of the lymphoma returning even after receiving high dose chemotherapy with stem cell transplantation. In order to improve the response and decrease the relapse rate, additional therapy may be used to kill the lymphoma cells by using antibodies both before and after the transplantation. Antibodies are protein made by white cells in our body to fight off infection and sometimes tumor. Rituxan (rituximab) is an antibody that is effective against your type of lymphoma. Researchers have reported that patients show an improved response and a lower chance of relapse when using rituximab with high dose chemotherapy with autologous stem cell transplantation. It is unknown how effective rituximab is in clearing persistence of minimal remaining disease in patients with follicular lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy-proven refractory CD20+ (cluster of differentiation antigen 20) Follicular lymphoma or transplant eligible mantle cell lymphoma in CR1 (complete remission 1) or later.
* Patients must be transplant eligible per KUCC BMT SOP (Kansas University Cancer Center Bone Marrow Transplant Standard Operation Procedures) with chemo-sensitive/marrow negative disease.
* Patients planning to harvest and hold may also be included as long as above criteria are met.

Exclusion Criteria:

* Pregnancy
* Zubrod performance status greater than 2
* Life expectancy is severely limited by concomitant illness.
* Uncontrolled arrhythmias or symptomatic cardiac disease precluding transplantation
* Symptomatic pulmonary disease precluding transplantation
* Serum creatinine greater than 1.8 mg/dL
* Serum bilirubin greater than 2 X upper limit of normal, SGPT (serum glutamate pyruvate transaminase) greater than 3 times upper limit of normal
* Evidence of chronic active hepatitis or cirrhosis
* Unable to sign informed consent.
* Allergy to Rituximab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-02; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Siddhartha Ganguly, MD, Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kansas Medical Center, Westwood Campus, Kansas City, Kansas

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab: Rituximab: 375 MG/M2 given IV weekly x 4-8 doses.
Period: Overall Study
Arm/Group | Rituximab
Started | 19
Completed | 14
Not Completed | 5
Not completed — Was not transplanted | 5

BASELINE CHARACTERISTICS:
Arm/Group | Rituximab
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Rate of PCR Negativity
Description: Number of participants that are tumor free by PCR (Polymerase Chain Reaction) analysis post-transplant.
Time Frame: up to 7 days
Population: 21 patients were initially enrolled; 2 were withdrawn after signing informed consent per physician decision. Of the remaining 19: 5 did not have harvestable stem cells; 14 completed stem cell collection and PCR evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab
Number analyzed (Participants) | 14
Participants | 14

2. Secondary Outcome: Progression Free Survival (PFS) and Overall Survival (OS)
Description: Response will be determined by Response Evaluation Criteria in Solid Tumors (RECIST v1.0) criteria where applicable and/or biopsy proven relapse/progression of disease.
Time Frame: up to 60 months
Population: Of the 14 patients that had harvestable cells, 3 chose to delay transplant. The remaining 11 patients underwent Autologous stem cell transplantation (Auto-SCT).
Measure: Median (Full Range); unit: months
Arm/Group | Rituximab
Number analyzed (Participants) | 11
months
  PFS in FL: number analyzed (Participants) | 7
  PFS in FL | 24 [9 to 60]
  OS in FL: number analyzed (Participants) | 7
  OS in FL | 36 [24 to 60]
  PFS in ML: number analyzed (Participants) | 4
  PFS in ML | 36 [24 to 48]
  OS in ML: number analyzed (Participants) | 4
  OS in ML | 48 [24 to 60]

ADVERSE EVENTS:
Time Frame: 1 year post-transplant or post-harvest
Arm/Group | Rituximab
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 1/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab (N=19)
Thrombosis/thrombus/embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes